CLINICAL TRIAL: NCT03640494
Title: Bedside Optical Retinal Assessment of Hypoxic Ischemic Encephalopathy in Infants
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00100417; 1R21EY029384 (NIH)
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-02

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Optical Coherence Tomography; Newborn; Infant
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates with a clinical HIE diagnosis: 48 neonates with a clinical diagnosis of HIE will be recruited from the patient populations of Duke University Health System and the University of Utah. All subject will have bedside optical coherence tomography (OCT) imaging performed at various time points while in the intensive care nursery.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — This is an observational study in which subjects will be imaged with optical coherence tomography (OCT). OCT systems are optical imaging technology that allow non-contact imaging of the microanatomy of the retina, optic nerve head and retinal blood vessels. The OCT devices are held above (and do not touch) the eye. Unlike visible light from many examination devices, the infrared OCT beam is barely visible to the human eye as it sweeps across the retina. Thus the infant is not disturbed by the light.

SUMMARY:
The purpose of this study is to develop a novel noninvasive bedside optical coherence tomography (OCT) imaging technique in newborn infants with HIE that improves our ability to assess the range of retinal effects from HIE and to diagnose and monitor treatments of HIE.

ELIGIBILITY:
Inclusion Criteria:

Infants are eligible if:

* Admitted to the intensive care nursery, outborn or inborn, with a clinical diagnosis of HIE; and with the approval of the neonatologist
* A parent or legal guardian provides written informed consent

Exclusion Criteria:

Potentially eligible infants will be excluded if:

• Congenital or chromosomal anomaly that has a profound impact on brain or eye development (e.g. anencephaly, congenital cataract or Peter's anomaly) and infants for whom there has been a clinical decision to limit life support.

Max Age: 20 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Forty-eight participants with a clinical diagnosis of hypoxic ischemic encephalopathy will be recruited and consented into this study from the patient populations of Duke University and the University of Utah neonatal intensive care nurseries.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Retinal injury morphologies on optical coherence tomography | birth to 10 days
  Composite injury score from presence or absence of 5 morphologies on optical coherence tomography: 1) cystoid spaces,2) ganglion cell layer abnormality, 3) paracentral acute middle maculopathy, 4) hemorrhages, 5) photoreceptor ellipsoid zone at the fovea
Retinal nerve fiber layer thickness on optical coherence tomography | birth to 10 days
  Deviation in the retinal nerve fiber layer thickness in the papillomacular bundle: 0 to 150 microns
Inner macular layer thickness on optical coherence tomography | birth to 10 days
  Deviation in the thickness from internal limiting membrane to outer plexiform layer across the macula (500, 1000 and 2000μm from the fovea): 0 to 500 microns
Clinical hypoxic ischemic encephalopathy score | birth to 6 hours
  hypoxic ischemic encephalopathy clinical score, within the first 6 hours of life, based on the modified Sarnat staging scale: mild, moderate or severe
MRI brain injury score | from 4 to 14 days after birth
  MRI scoring: global score of overall injury [0-138] characterized as mild [0-11], moderate [12-32], or severe [>32].

SECONDARY OUTCOMES:
Total macular layer thickness on optical coherence tomography | birth to 9 weeks
  Deviation in total retinal thickness across macula (500, 1000 and 2000μm from the fovea): 0 to 500 microns
Center foveal thickness | birth to 9 weeks
  Deviation in retinal thickness at the foveal center
Center ellipsoid zone thickness | birth to 9 weeks
  Deviation in retinal thickness at the foveal center: 0 to 100 microns
pattern of MRI injury | from 4 to 14 days after birth
  Patterns of injury characterized descriptively as white matter, focal cortical, deep nuclear brain matter, or global based on the scoring methods of Bednadrek N et al.
Choroidal thickness on optical coherence tomography | birth to 9 weeks
  Deviation in choroidal thickness across macula(500, 1000 and 2000μm from the fovea): 20 to 800 microns
Optic nerve head morphology | birth to 9 weeks
  optic nerve head elevation and cup as a composite morphology: normal, excavated, elevated, bowing of retinal pigment epithelium
thickness of macular nerve fiber layer | birth to 9 weeks
  Deviation in nerve fiber layer thickness across macula(500, 1000 and 2000μm from the fovea): 0 to 100 microns
thickness of macular ganglion cell layer | birth to 9 weeks
  Deviation in ganglion cell layer thickness across macula(500, 1000 and 2000μm from the fovea): 0 to 200 microns
thickness of inner nuclear layer | birth to 9 weeks
  Deviation in total retinal thickness across macula (500, 1000 and 2000μm from the fovea): 0 to 400 microns
thickness of inner plexiform layer | birth to 9 weeks
  Deviation in inner plexiform layer thickness across macula (500, 1000 and 2000μm from the fovea): 0 to 100 microns
thickness of photoreceptor layer | birth to 9 weeks
  Deviation in total retinal thickness across macula(500, 1000 and 2000μm from the fovea): 0 to 200 microns
Longitudinal change in retinal injury morphologies on optical coherence tomography | birth to 9 weeks
  Composite injury score from presence or absence of 5 morphologies on optical coherence tomography: 1) cystoid spaces,2) ganglion cell layer abnormality, 3) paracentral acute middle maculopathy, 4) hemorrhages, 5) photoreceptor ellipsoid zone at the fovea
Longitudinal change in retinal nerve fiber layer thickness on optical coherence tomography | birth to 9 weeks
  Deviation in the retinal nerve fiber layer thickness in the papillomacular bundle: 0 to 150 microns
Longitudinal change in inner macular layer thickness on optical coherence tomography | birth to 9 weeks
  Deviation in the thickness from internal limiting membrane to outer plexiform layer across the macula (500, 1000 and 2000μm from the fovea): 0 to 500 microns
Late clinical hypoxic ischemic encephalopathy score | 1 to 8 days
  Composite hypoxic ischemic encephalopathy severity score based on: examination after rewarming, early feeding behavior score, seizure score and electroencephalogram score

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Toth, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Health System, Durham, North Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran-Viet D, Wong BM, Mangalesh S, Maldonado R, Cotten CM, Toth CA. HANDHELD SPECTRAL DOMAIN OPTICAL COHERENCE TOMOGRAPHY IMAGING THROUGH THE UNDILATED PUPIL IN INFANTS BORN PRETERM OR WITH HYPOXIC INJURY OR HYDROCEPHALUS. Retina. 2018 Aug;38(8):1588-1594. doi: 10.1097/IAE.0000000000001735. PMID 28570486
- [Result] Mangalesh S, Tran-Viet D, Pizoli C, Tai V, El-Dairi MA, Chen X, Viehland C, Edwards L, Finkle J, Freedman SF, Toth CA. Subclinical Retinal versus Brain Findings in Infants with Hypoxic Ischemic Encephalopathy. Graefes Arch Clin Exp Ophthalmol. 2020 Sep;258(9):2039-2049. doi: 10.1007/s00417-020-04738-0. Epub 2020 May 29. PMID 32472201